CLINICAL TRIAL: NCT03659474
Title: Different Cryotherapy Techniques for Skin Surface Temperature, Agility and Balance of Active Youth: Analysis Between Ice Pack, Cryoimmersion and Game Ready®
Brief Title: Different Cryotherapy Techniques for Skin Surface Temperature, Agility and Balance of Active Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Cryotherapy Techniques
Record Dates: First submitted 2018-02-16; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-04

CONDITIONS: Temperature
Keywords: skin temperature; postural control; ankle
MeSH Terms: interventions — Immersion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cryotherapy by compression (Experimental): maximum dynamic intermittent compression, programmed to maintain a temperature at 1 ° C
  Interventions: Other: compression
- ice pack (Experimental): the ankle joint was surrounded by three plastic bags containing crushed ice.
  Interventions: Other: ice pack
- cold water immersion (Experimental): articulation of the ankle submerged in cold water at approximately 10 ° C, being controlled by the thermal camera.
  Interventions: Other: immersion

INTERVENTIONS:
Other: compression — compression by Game Ready
  Arms: cryotherapy by compression
Other: ice pack — cryotherapy for ice pack
  Arms: ice pack
Other: immersion — immersion therapy
  Arms: cold water immersion

SUMMARY:
Different techniques of cryotherapy application present divergent responses. The objective was to establish differences between methods of application of ankle cryotherapy on skin surface temperature (TSP), agility and balance. The sample consisted of 20 healthy and active young men, 10 men and 10 women, with 21.4 (1.9) years. Initially, all performed the Modified Star Excursion Balance Test, Side Hop Test, and TSP collection of the lateral ankle region by digital thermography. After that, the application of the cryotherapy techniques - ice pack (PG), cold water immersion (LAI) and cryotherapy + compression by Game Ready® (CCGR), all for 20 minutes (') was randomized. The tests and TSP were reassessed in the immediate post-10'', 20'' and 30 'post. After three and six days, the other application forms were reassessed. Thus, the participants were randomly assigned to the three forms of cryotherapy.

DETAILED DESCRIPTION:
The present study is a longitudinal, randomized clinical trial with a composite sample of physically active individuals, 10 male volunteers and 10 female volunteers, with no history of lower limb injuries and pain complaints at the time collection. The collection will started after the signing of the free and informed consent form. The study was approved by the Research Ethics Committee of the State University of Londrina (UEL), Londrina, Paraná (Resolution 466/2012).

The sample size was calculated using the Power and Sample Size software, with a 95% confidence interval, 5% alpha force and 90%, considering the raw data (mean ± SD) of the surface temperature in the study, "The Magnitude of Tissue Cooling During Cryotherapy With Varied Types of Compression ", where it presented 11.02 and 15.51 as mean, 4.34 of standard deviation and p <0.05. sample was composed of 20 individuals per group.

Initially, a pre-intervention evaluation will performed, where the superficial skin temperature of the ankle region will collected from the participants with a professional Flir C2® thermal camera and two functional tests will be performed: Y test and Side Hop Test (SHT) . After the baseline assessment the participants performed will walk at a constant and comfortable pace.

Immediately after walking, subjects will referred to one of three cryotherapy techniques to be tested: Game Ready® cryotherapy (CGR), ice pack cryotherapy (PG) or cold water ankle immersion (IAF).

For the CGR group, maximum dynamic intermittent compression will used, programmed to maintain a temperature at 1 ° C. In the PG group, the ankle joint will surrounded by three plastic bags containing crushed ice. The IAF group will remain with the ankle joint submerged in cold water at approximately 10 ° C, being controlled by the thermal camera. All treatments were performed for 20 minutes.

The same temperature assessment will performed immediately after 10 minutes, 20 minutes, 30 minutes and 60 minutes after cryotherapy, while the functional tests were re-evaluated immediately, 10, 20 and 30 minutes. The participants will attend for data collection on three distinct days, randomizing one of three interventions each day.

For the performance of the functional tests, the order of onset will randomized. The SHT will analyze the agility of the participant, submitting it in unipodal support with the dominant lower limb without shoes, performing 10 distal mid-lateral jumps about thirty centimeters, as fast as possible, being performed three times. The balance will analyzed through the Y test, with the barefoot participant positioned the dominant foot, at the intersection between all diagonals, so that the malleolar line would be in the center of them, and with the other foot the participants pushed a small, light box as far as he can without removing his support foot. Statistical analysis will be performed using SPSS software version 2.2, and the level of significance was set at 5%. It will used and test and Shapiro Wilk to test the normality of the data. From this, the ANOVA test will be used to compare study groups and moments studied.

ELIGIBILITY:
Inclusion Criteria:

* physically active
* no history of lower limb injuries
* no complaints of pain at the time of collection

Exclusion Criteria:

* sedentary
* injury or ankle surgery

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Change in skin surface temperature after intervention | pre-intervention, Immediately after, post 10, 20 and 30 minutes
  evaluated by professional thermal camera Flir C2®

SECONDARY OUTCOMES:
Change in agility after intervention | pre-intervention, Immediately after, post 10, 20 and 30 minutes
  evaluated by Side Hop Test
Change in postural control after intervention | pre-intervention, Immediately after, post 10, 20 and 30 minutes
  evaluated by Y test

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Macedo, Principal Investigator — State University of Londrina
Locations (1):
- Christiane Macedo, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tomchuk D, Rubley MD, Holcomb WR, Guadagnoli M, Tarno JM. The magnitude of tissue cooling during cryotherapy with varied types of compression. J Athl Train. 2010 May-Jun;45(3):230-7. doi: 10.4085/1062-6050-45.3.230. PMID 20446835